CLINICAL TRIAL: NCT01862367
Title: Use of rFXIII in Treatment of Congenital FXIII Deficiency, a Prospective Multi-centre Observational Study
Acronym: mentor™6
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1841-3868; U1111-1131-1558 (Other: WHO); ENCEPP/SDPP/3687 (Registry Identifier: EU PAS)
Record Dates: First submitted 2013-05-21; First posted 2013-05-24 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency
MeSH Terms: interventions — recombinant factor XIII-A2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rFXIII
  Interventions: Drug: catridecacog

INTERVENTIONS:
Drug: catridecacog — No treatment given. All patients enrolled in this observational study will receive their medication through usual commercial channels.
  Other Names: recombinant factor XIII

SUMMARY:
This study is conducted globally. The aim of this observational study is to investigate the incidence of specific adverse drug reactions associated with the use of recombinant factor XIII (NovoThirteen®) in patients with congenital FXIII A-subunit deficiency (congenital FXIII deficiency), comprising FXIII antibodies, allergic reactions, embolic and thrombotic events and lack of therapeutic effect.

The study will aim at observing all patients exposed to NovoThirteen® in the EU, and additional patients from selected non-EU countries. Recombinant FXIII (rFXIII) is registered in EU and Switzerland as NovoThirteen® and in Canada as Tretten®.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. (Study-related activities are any procedure related to recording of data according to the protocol)
* Able and willing to provide signed informed consent (or patient's legally acceptable representative (LAR) consent, if applicable), as required by local ethics committee, governmental or regulatory authorities
* Congenital FXIII A-subunit deficiency
* Actual or planned exposure to rFXIII

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational study will enroll patients with congenital FXIII A-subunit deficiency for whom the decision to treat with rFXIII has been made and who are willing to provide informed consent (or patient's legally acceptable representative (LAR) consent, if applicable).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Adverse drug reactions in patients with congenital FXIII A-subunit deficiency treated with rFXIII,comprising FXIII antibodies, allergic reactions, embolic and thrombotic events and lack of effect collected | During study period up to 6 years

SECONDARY OUTCOMES:
All serious adverse events collected | During study period up to 6 years
All medical events of special interest collected | During study period up to 6 years
All medication errors and near medication errors collected | During study period up to 6 years
Use of rFXIII in patients with congenital FXIII A-subunit deficiency also for other uses than for prophylactic treatment collected | During study period up to 6 years
Frequency of bleeding episodes collected | During study period up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- United States (7):
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
- Canada (2):
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Toronto, Ontario
- Novo Nordisk Investigational Site, Debrecen, Hungary
- Italy (2):
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Genova
- Spain (4):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Tortosa
- Novo Nordisk Investigational Site, Aberdeen, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com